CLINICAL TRIAL: NCT07175025
Title: The New Empowerment After eXposure to Trauma (NEXT) Study
Acronym: NEXT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michelle L. Miller, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23HD115845 (NIH); K23HD115845 (NIH)
Record Dates: First submitted 2025-09-03; First posted 2025-09-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: PTSD - Post Traumatic Stress Disorder; PTSD (Childbirth-Related)
Keywords: Pregnancy; Postpartum Period; Narrative Exposure Therapy; Post-Traumatic Stress Disorder; Brief interventions
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Potential participants will be screened to determine eligibility. If interested and eligible, informed consent will be obtained prior to beginning the study. After signing consent, participants will be asked to complete a self-report baseline assessment. After collection of baseline data, participants will be randomized 1:1 to the NET intervention or usual care group. Block randomization will be used with computer-generated randomization lists provided by the study statistician. All participants will be asked to complete self-report assessments at standard intervention assessment time points: Time 1 (0 weeks; baseline) Time 2 (12 weeks; post-intervention) and Time 3 (24 weeks; 3-month follow-up). Qualitative feedback will be gathered at Time 3, after other data collection is complete. Recruitment procedures, eligibility determination, and assessments will be identical for both groups. Study participation will last 24 weeks, starting at Time 1 (Week 0).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants will complete a brief Narrative Exposure Therapy (NET) intervention. NET is a potent exposure-based intervention that is fully manualized, short-term, and developed for individuals with multiple traumas. NET is effective in as little as four sessions and can be completed virtually. NET involves four parts: 1) psychoeducation on trauma exposure and PTSD, 2) laying the Lifeline (constructing a life events inventory, including meaningful events and trauma exposures), 3) exposure sessions (retelling of a traumatic event while constructing the trauma narrative in the context of the life course), and 4) reading of the full written narrative, written by the study therapist after each exposure.
  Interventions: Behavioral: Narrative Exposure Therapy (NET)
- Usual Care Group (No Intervention): This group will receive usual care for physical and mental health concerns during pregnancy and the postpartum period. Participation in the usual care group will consist of symptom monitoring (study staff) and participant's primary care/obstetric care for all other concerns. After enrollment in the study, the research assistant will have a structured 10-15 call/visit with usual care group participants to assess existing psychosocial support/health providers and provide a list of mental health services across IUSM and the state of Indiana/perinatal supports. They will encourage participants to follow-up with their primary care/obstetric care provider/community organizations for more help if needed. All usual care group participants will be offered the NET intervention after study assessments have been collected.

INTERVENTIONS:
Behavioral: Narrative Exposure Therapy (NET) — Narrative Exposure Therapy (NET) is the PTSD intervention for the treatment group.
  Arms: Treatment Group

SUMMARY:
The NEXT Study is a randomized controlled pilot examining the feasibility and acceptability of a revised perinatal PTSD protocol. This study will randomize perinatal participants with PTSD to receive NET (n=45); treatment group) and will be compared to perinatal women randomized to usual care (n=45; comparator group). The overall objective of this project is to determine the most feasible and acceptable protocol for a brief virtual perinatal PTSD intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* able to read and speak English
* diagnosis of probable PTSD as determined by the PTSD Checklist for DSM-5 (PCL-5)
* pregnant or postpartum (delivered within 16 weeks) at the time of the eligibility screen Exclusion criteria
* current severe suicide risk
* current psychotic or manic symptoms
* cognitive impairment
* concurrent trauma-focused psychotherapy
* medical advice limiting participation in exposure therapy
* current legal actions related to trauma
* does not meet criteria for PTSD
* not pregnant or delivered more than 12 weeks after timing of eligibility screening

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Tracking | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  The investigators will determine feasibility by enrollment (≥75% of potential participants enroll), treatment adherence (≥80% of treatment group complete 5/6 NET sessions), assessment completion/each time point (≥75% of sample), and study completion (≥75% of sample).
Acceptability | Post-intervention time period (12 weeks post-baseline)
  The Triple P-Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), & Feasibility of Intervention Measure (FIM) scales will be used to assess overall acceptability of the NEXT protocol
Perinatal NET Protocol Acceptability Questionnaire (PNPAQ) | Post-intervention time period (12 weeks post-baseline) for the NET treatment group
  A 20-item study-specific measure used to assess various PNET protocol components as well as 10 exploratory questions on acceptability of potential future protocol elements (e.g., collection biomarkers, in person v. virtual).

SECONDARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | *Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline). *Weekly to biweekly administration across 12 week intervention period
  Self-report assessment of PTSD symptoms in response to a traumatic event in past week or past month
Edinburgh Postnatal Depression Scale (EPDS) | *Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline). *Weekly to biweekly administration across 12 week intervention period
  Self-report assessment of depressive symptoms in the perinatal period, including suicidality.
Life Events Checklist (LEC) | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  Used to self-report traumatic events over the lifetime at start of study as well as any new traumas experienced during treatment period.
Perinatal Quality of Life | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  Mother-Generated Index (MGI) will be used to assess valued life domains by specifying up to eight areas of their lives which have been affected by being pregnant/ giving birth to a baby, assessing how the participant felt about this area over the previous month, and describing the domains most important to her.

OTHER OUTCOMES:
Parental Stress Scale (PSS) | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  Exploratory self-report measure that assesses participants' feelings about their parenting role
Treatment Tracking | *Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline) *Weekly to biweekly across 12 week intervention time period
  A brief study-specific measure to assess changes to medication doses and/or psychotherapy
Perinatal Life Events Checklist | Baseline and follow-up (24 weeks post-baseline)
  Exploratory study specific self-report measure used to assess potentially traumatic events that occur during pregnancy and the postpartum period.
Posttraumatic Growth Inventory (PGI) | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  A self-report measure assessing to assess post-trauma growth and self-improvement a person undergoes.
Centrality of Event (CE) | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  This 7-item measure assesses how central a traumatic event is to a participant's identity and life story and if that changes with intervention.
Social Isolation | Baseline, post-intervention time period (12 weeks post-baseline), and follow-up (24 weeks post-baseline)
  The UCLA 3-item Social Isolation scale will be used to assess loneliness and social isolation, a predictor of maternal health.
Therapist Alliance | *Week 4 of intervention period *Post-intervention time period (12 weeks post-baseline) for the NET treatment group
  The Working Alliance Inventory-Short-Form (WAI-SF) will be used to assess how participant feels about fit with study therapist assigned to them at mid- and end of treatment.
Eligibility | Eligibility screening that occurs before baseline assessment
  The Mood Disorder Questionnaire (MDQ) will be used to screen for mania symptoms and exclude ineligible individuals
Eligibility | Eligibility screening that occurs before baseline assessment
  The Columbia Suicide Severity Screening will be used to assess for higher levels of suicidality and used to exclude individuals that have too high of suicidality levels to be cared for through a brief, virtual PTSD intervention
Eligibility | Eligibility screening that occurs before baseline assessment
  The Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders (DIAMOND) screener for psychosis symptoms will be used to exclude individuals that endorse psychosis symptoms and thus need a higher level of care than can be offered through a brief, virtual PTSD intervention

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L. Miller, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share the study protocol, Statistical Analysis Plan (SAP), and Informed Consent Form (ICF)
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The Study Protocol and SAP will be pre-registered and available at the start of the trial (9/15/25). The Informed Consent form will be approved by the Institution IRB prior to the start of the trial and available by request. There is not a specified end date for these materials.
Access Criteria: The study team currently has access to all documents and the Study Protocol and SAP are available through the OSF preregistration website.

REFERENCES:
- [Background] Kays MB, Wack MF, Smith DW, Denys GA. Azithromycin treatment failure in community-acquired pneumonia caused by Streptococcus pneumoniae resistant to macrolides by a 23S rRNA mutation. Diagn Microbiol Infect Dis. 2002 Jun;43(2):163-5. doi: 10.1016/s0732-8893(02)00379-6. PMID 12088625
- [Background] Stevens NR, Miller ML, Soibatian C, Otwell C, Rufa AK, Meyer DJ, Shalowitz MU. Exposure therapy for PTSD during pregnancy: a feasibility, acceptability, and case series study of Narrative Exposure Therapy (NET). BMC Psychol. 2020 Dec 9;8(1):130. doi: 10.1186/s40359-020-00503-4. PMID 33298159